CLINICAL TRIAL: NCT07106502
Title: Learning to Palpate the Child's Testicles Using Simulation
Acronym: PaTenSim
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC24_0256
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Testicular Positioning Anomalies; Cryptorchidism
Keywords: cryptorchidism; testicular palpation
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- mannequin simulation-based learning group (Experimental)
  Interventions: Procedure: testicular palpation training on a mannequin

INTERVENTIONS:
Procedure: testicular palpation training on a mannequin — Study of testicular palpation training on a mannequin on the ability to perform a testicular examination and diagnose testicular positioning abnormalities
  Arms: mannequin simulation-based learning group

SUMMARY:
Hypothesis is that better training of medical students in the examination of boy's external genitalia could improve the diagnosis of testicular position anomalies. To this end, investigators already have created a model to train testicle palpation and recognition of testicular position anomalies. So investigator set up a monocentric randomized controlled trial in wich the medical students will be randomized into 2 groups : a control group receiging only book-based theoretical instruction on the examination of the external genitalia and testicular position anomalies, and a mannequin group receibing, in addition to this conventionnal instruction, simulation training on the mannequin Medical students will then attend a consultation with a child whose reason for coming to the hospital is a testicular positioning anomaly. Students clinical examination will be scored by the consulting senior, and the final diagnosis retained by the student will be compared with that retained by the consulting senior. The aim is to show that medical students who have trained on this new model are better, in terms of clinical examination and diagnostic, than students in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Medical student who volunteers to take part in the study during their pediatric or pediatric surgery clerkship or at the simulation center

Exclusion Criteria:

* student non in pediatric intership or non in pediatric surgery intership or non at the simulation center intership
* Student with previous simulation training in the examination of the external genitalia of children

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of correct diagnoses | Baseline
  The primary outcome will be the rate of correct diagnoses made by the medical students compared with the diagnosis made by the consultant surgeon.

SECONDARY OUTCOMES:
clinical examination score from 0 to 20 | Baseline
  to assess the student's clinical skills and the quality of the physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Louise RENOULT, Study Chair — University Hospital of Angers

IPD SHARING:
Plan to Share IPD: Undecided